CLINICAL TRIAL: NCT04736966
Title: A Phase I Clinical Trial to Determine the Safety and Tolerability of Anti-IL23 Monoclonal Antibody, for the Treatment of Patients With Alcohol Associated Liver Disease
Brief Title: Guselkumab (Anti-IL 23 Monoclonal Antibody) for Alcohol Associated Liver Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Rohit Loomba, Professor of Medicine, University of California, San Diego
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Anti-IL23 Trial Phase 1
Record Dates: First submitted 2021-01-19; First posted 2021-02-03 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Alcoholic Liver Disease
MeSH Terms: conditions — Liver Diseases, Alcoholic | interventions — guselkumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Guselkumab 30mg (Experimental): Guselkumab administered by subcutaneous injection at Day 1 and Day 29
  Interventions: Drug: Guselkumab 30mg
- Guselkumab 70 mg (Experimental): Guselkumab administered by subcutaneous injection at Day 1 and Day 29
  Interventions: Drug: Guselkumab 70mg
- Guselkumab 100mg (Experimental): Guselkumab administered by subcutaneous injection at Day 1 and Day 29
  Interventions: Drug: Guselkumab 100mg

INTERVENTIONS:
Drug: Guselkumab 30mg — 30mg of Guselkumab administered by subcutaneous injection
  Other Names: Tremfya
  Arms: Guselkumab 30mg
Drug: Guselkumab 70mg — 70mg of Guselkumab administered by subcutaneous injection
  Other Names: Tremfya
  Arms: Guselkumab 70 mg
Drug: Guselkumab 100mg — 100mg of Guselkumab administered by subcutaneous injection
  Other Names: Tremfya
  Arms: Guselkumab 100mg

SUMMARY:
A Phase I clinical trial to determine the safety and tolerability of an anti-IL23 antibody for the treatment of patients with alcoholic liver disease

DETAILED DESCRIPTION:
This is a phase I study of guselkumab, a humanized anti-IL23 monoclonal antibody, for patients with alcoholic liver disease. This drug is approved for the use in psoriatic arthritis but not for alcoholic liver disease. The investigators will be using a standard 3+3 phase I dose escalation trial design, the dose levels will start from 30 mg, 70 mg and to 100 mg, a maximum total of 24 patients will be evaluable. In this study the investigators propose to establish safety of the product in those with alcoholic liver disease and efficacy (secondary endpoint) will be determined by biomarkers for liver inflammation and fibrosis surrogate biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent (either from patient or patient's legally acceptable representative)
2. Male or female patients 21 years of age or older with BMI ≥ 20 to ≤ 45 kg/m2
3. Patients with moderate alcohol use disorder (AUD) as defined by the AASLD Practice Guidance to have ≥ 4 symptoms out of 11:

   1. Alcohol is often taken in larger amounts and/or over a longer period than the patient intended.
   2. Persistent attempts or one or more unsuccessful efforts made to cut down or control alcohol use.
   3. A great deal of time is spent in activities necessary to obtain alcohol, use alcohol, or recover from effects.
   4. Craving or strong desire or urge to use alcohol
   5. Recurrent alcohol use resulting in a failure to fulfill major role obligations at work, school, or home.
   6. Continued alcohol use despite having persistent or recurrent social or interpersonal problem caused or exacerbated by the effects of the alcohol.
   7. Important social, occupational or recreational activities given up or reduced because of alcohol use.
   8. Recurrent alcohol use in situations in which it is physically hazardous.
   9. Alcohol use is continued despite knowledge of having a persistent or recurrent physical or psychological problem that is likely to have been caused or exacerbated by the alcohol.
   10. Tolerance, as defined by either of the following:

   <!-- -->

   1. Markedly increased amounts of the alcohol in order to achieve intoxication or desired effect
   2. Markedly diminished effect with continued use of the same amount

   k. Withdrawal, as manifested by either of the following:
   1. The characteristic alcohol withdrawal syndrome or
   2. Alcohol (or a closely related substance) is taken to relieve or avoid withdrawal symptoms
4. Evidence of end-organ damage to the liver as defined by

   a. MRI-PDFF ≥ 8% suggestive of significant hepatic accumulation of triglyceride within 3 months of screening; if patients cannot get an MRI, CAP ≥ 300dB/m
5. Consumed alcohol within 12 weeks of entry into the study, AND

   a. AST and ALT less than 200 U/L AND
6. No evidence of active infection as determined by the investigator.
7. Women of child-bearing potential (defined as females who are not surgically sterile or who are not over the age of 52 and amenorrheic for at least 12 months) must utilize appropriate birth control throughout the study duration. Acceptable methods that may be used are abstinence, birth control pills ("The Pill") or patch, diaphragm, intrauterine device (IUD/ coil), vaginal ring, condom, surgical sterilization or progestin implant or injection, or sexual activity limited to a sterile (e.g., vasectomized) male partner.
8. Male patients must agree to use a medically acceptable method of contraception/birth control throughout the study duration.

Exclusion Criteria:

1. History or evidence of other or concomitant cause(s) of liver disease as a result of:

   1. Autoimmune liver disease
   2. Wilson disease (ceruloplasmin levels < 10 mcg/L)
   3. Vascular liver disease
   4. Drug induced liver disease
   5. Surface antigen positive hepatitis B (HBsAg+). Note: patients with isolated core antibody (HBcAb) are not excluded.
   6. Acute hepatitis A
   7. Acute HCV or chronic hepatitis C with a history of decompensated cirrhosis. (Note: patients with stable chronic Hep C Virus (HCV) or successfully treated HCV are not excluded. Anti-HBc antibody positive patients will be given a prophylaxis with entecavir 0.5mg PO once daily, starting one week prior to start of guselkumab to 6 months after the last dose of guselkumab)
2. Noninvasive criteria to exclude cirrhosis:

   1. MRE ≥ 3.63 kPa; if MRE not available, VCTE ≥ 16 kPa
   2. FIB-4 ≥ 2.67
   3. Imaging evidence of varices, splenomegaly, ascites, or shrunken cirrhotic liver
3. Co-infection with human immunodeficiency virus (HIV)
4. History or evidence of positive Urine Drug Screen (amphetamines, barbiturates, benzodiazepines, cocaine and opiates) except THC and legal prescription medications.
5. Any active malignancies other than curatively treated skin cancer (basal cell or squamous cell carcinomas) or any other malignancy diagnosed within the last five years
6. History or evidence of active tuberculosis
7. Positive Quantiferon test
8. Significant systemic or major illness other than liver disease, including coronary artery disease, cerebrovascular disease, pulmonary disease, renal failure, serious psychiatric disease, that, in the opinion of the Investigator would preclude the patient from participating in and completing the study
9. Patients requiring the use of vasopressors or inotropic support.
10. Any patient that has received any investigational drug within 30 days of dosing or who is scheduled to receive another investigational drug at any time during the study
11. Patients who are taking drug products that are primarily the substrates of CYP2C8, such as chloroquine, paclitaxel, rosiglitazone, repaglinide
12. If female, known pregnancy, or has a positive serum pregnancy test, or is lactating/breastfeeding
13. Serum creatinine > 1.5 mg/dL
14. Patients who have had organ transplantation (such as liver, kidney, lung, heart, bone marrow, or stem cell etc.), other than cornea transplant
15. Presence of cirrhosis on imaging or any of following lab parameters:

    1. Albumin < 3.7 g/dL
    2. Direct bilirubin > 0.5 mg/dl unless due to Gilbert's syndrome
    3. Platelets < 140K
    4. INR > 1.3
16. Presence of any features of portal hypertension such as ascites, history of ascites or varices, or encephalopathy
17. Previous use of guselkumab ( or another IL-23 inhibitors) or hypersentivity to guselkumab
18. Previous history of skin cancers in the last one year
19. Previous history of breast or prostate cancer or any cancer within the last 5 years

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Assess the safety and tolerability of Guselkumab | 48 Weeks
  Incidence of treatment-emergent adverse events: Outcome measures will include incidence of treatment-emergent adverse events and the proportion of subjects prematurely withdrawn from the study due to adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Loomba, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No